CLINICAL TRIAL: NCT01980303
Title: An Open-label, Single-Dose Study to Assess the Pharmacokinetics, Safety and Tolerability of Intranasally Administered Esketamine in Healthy Japanese and Caucasian Subjects
Brief Title: A Study to Assess the Pharmacokinetics of Intranasally Administered Esketamine in Healthy Japanese and Caucasian Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR101101; ESKETINTRD1002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Healthy Volunteers
Keywords: Healthy; Japanese; Caucasian; Anesthetics; Intranasal; Esketamine; Pharmacokinetics
MeSH Terms: interventions — Esketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1: Treatment A (Experimental): Japanese participants will receive 1 spray of esketamine solution in each nostril (total dose: 28 mg).
  Interventions: Drug: Esketamine
- Cohort 1: Treatment B (Experimental): Japanese participants will receive 1 spray of esketamine solution in each nostril at time 0 and 5 minutes (total dose: 56 mg).
  Interventions: Drug: Esketamine
- Cohort 1: Treatment C (Experimental): Japanese participants will receive 1 spray of esketamine solution in each nostril at time 0, 5, and 10 minutes (total dose: 84 mg).
  Interventions: Drug: Esketamine
- Cohort 2: Treatment A (Experimental): Caucasian participants will receive 1 spray of esketamine solution in each nostril (total dose: 28 mg).
  Interventions: Drug: Esketamine
- Cohort 2: Treatment B (Experimental): Caucasian participants will receive 1 spray of esketamine solution in each nostril at time 0 and 5 minutes (total dose: 56 mg).
  Interventions: Drug: Esketamine
- Cohort 2: Treatment C (Experimental): Caucasian participants will receive 1 spray of esketamine solution in each nostril at time 0, 5 and 10 minutes (total dose: 84 mg).
  Interventions: Drug: Esketamine

INTERVENTIONS:
Drug: Esketamine — Fourteen percent esketamine solution (14 mg of esketamine per 100 microliter) will be administered intranasally by nasal spray pump.

SUMMARY:
The purpose of this Phase 1 study is to characterize the pharmacokinetic profile (what the body does to the medication) of esketamine when given by the intranasal route (through the nose) to healthy adult Japanese and Caucasian participants.

DETAILED DESCRIPTION:
This is an open-label single-center study with 2 cohorts (groups). The study will consist of a screening phase, a treatment phase, and a follow-up visit (9 to 13 days after the last dose of the study drug). During the screening phase, participants will be evaluated to determine if they meet the study eligibility criteria. A target of 14 healthy Japanese and 14 healthy Caucasian adult participants (20 to 55 years of age inclusive) will be enrolled in Cohort 1 and Cohort 2, respectively.

The participants in each cohort will self-administer each of the 3 different single-dose regimens of intranasal esketamine (Treatments A, B, and C) over the 3 treatment periods (ie, 1 treatment per period) in an open-label manner (both the investigator and the participant knows which intervention the participant receives). The participants will be randomly (like the toss of a coin) assigned to receive Treatment A and Treatment B in the first two periods (ie, Treatment A in Period 1 and Treatment B in Period 2, or the reverse order). All participants will receive Treatment C in Period 3. The regimens differ in the number of sprays to achieve the total dose and the total esketamine dose administered.

Safety and tolerability will be evaluated throughout the study and will include assessment of adverse events, targeted nasal examinations, laboratory tests, electrocardiogram, physical examination, pulse oximetery, and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese (Cohort 1) or Caucasian (Cohort 2) man or woman, between 20 to 55 years of age
* Resided outside of Japan for no more than 5 years and have parents and maternal and paternal grandparents who are of Japanese ethnicity
* Blood pressure (after the participant is in the supine position for 5 minutes) between 90 and 145 mmHg systolic, inclusive, and no higher than 90 mmHg diastolic
* A 12-lead electrocardiogram consistent with normal cardiac conduction and function
* Smokes no more than 10 cigarettes, or 2 cigars, or 2 pipes of tobacco per day for at least 6 months before first study drug administration
* Comfortable with self-administration of intranasal medication and able to follow instructions provided

Exclusion criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease; hematologic disease; coagulation disorders (including any abnormal bleeding or blood dyscrasias); hypertension or vascular disorders; significant pulmonary disease, including any bronchospastic respiratory disease; diabetes mellitus; renal or hepatic insufficiency; thyroid disease; neurologic or psychiatric disease, infection; kidney/urinary tract disturbances; sleep apnea, or myasthenia gravis, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening or at admission to the study center
* Anatomical or medical conditions that may impede delivery or absorption of study medication
* Has an abnormal or deviated nasal septum with any 1 or more of the following symptoms: blockage of 1 or both nostrils, nasal congestion (especially 1-sided), frequent nosebleeds, frequent sinus infections, noisy breathing during sleep, and at times has facial pain, headaches, and postnasal drip
* Has a current diagnosis of a psychotic disorder, bipolar disorder, mental retardation, or borderline personality disorders; mood disorder with postpartum onset, somatoform disorders, fibromyalgia, or chronic fatigue syndrome; generalized anxiety disorder, panic disorder, obsessive compulsive disorder, posttraumatic stress disorder, anorexia nervosa, or bulimia nervosa

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2013-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration during a dosing interval (Cmax) of esketamine and noresketamine | Predose, 7 minutes, 12 minutes, 22 minutes, 32 minutes, 40 minutes, 50 minutes, 1 hour, 1.25 hours, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 9 hours, 12 hours, 18 hours, 24 hours
Time to reach the maximum plasma concentration (tmax) of esketamine and noresketamine | Predose, 7 minutes, 12 minutes, 22 minutes, 32 minutes, 40 minutes, 50 minutes, 1 hour, 1.25 hours, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 9 hours, 12 hours, 18 hours, 24 hours
Area under the plasma concentration-time curve from Time 0 to time of the last quantifiable concentration of esketamine and noresketamine | Predose, 7 minutes, 12 minutes, 22 minutes, 32 minutes, 40 minutes, 50 minutes, 1 hour, 1.25 hours, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 9 hours, 12 hours, 18 hours, 24 hours
Elimination half-life of esketamine and noreskatamine | Predose, 7 minutes, 12 minutes, 22 minutes, 32 minutes, 40 minutes, 50 minutes, 1 hour, 1.25 hours, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 9 hours, 12 hours, 18 hours, 24 hours
Area under the plasma concentration-time curve from time 0 to infinite time in which Clast is the last observed quantifiable concentration of esketamine and noresketamine | Predose, 7 minutes, 12 minutes, 22 minutes, 32 minutes, 40 minutes, 50 minutes, 1 hour, 1.25 hours, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 9 hours, 12 hours, 18 hours, 24 hours

SECONDARY OUTCOMES:
The number of volunteers who experience adverse events as a measure of safety and tolerability. | Up to 71 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Cypress, California, United States

REFERENCES:
- [Derived] Perez-Ruixo C, Rossenu S, Zannikos P, Nandy P, Singh J, Drevets WC, Perez-Ruixo JJ. Population Pharmacokinetics of Esketamine Nasal Spray and its Metabolite Noresketamine in Healthy Subjects and Patients with Treatment-Resistant Depression. Clin Pharmacokinet. 2021 Apr;60(4):501-516. doi: 10.1007/s40262-020-00953-4. Epub 2020 Oct 31. PMID 33128208